CLINICAL TRIAL: NCT00875433
Title: Phase II Open Label Trial to Assess the Efficacy and the Impact on QTcF of Continuous Oral BIBW 2992 at a Daily Dose of 50mg in Patients With Relapsed or Refractory Solid Tumours Including Patients With Brain Metastases and Those With Glioblastoma Not Amenable to Other Therapy
Brief Title: Afatinib (BIBW 2992) QTcF Trial in Patients With Relapsed or Refractory Solid Tumours
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.24; 2008-006288-36 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Results first posted 2013-11-13 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-10

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib

ARMS (1):
- Monotherapy (Experimental): BIBW 2992 high dose, once daily, continuous, monotherapy
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992 — patients to receive continuous oral daily dosing of BIBW 2992

SUMMARY:
A phase II trial to assess the impact of afatinib (BIBW 2992) on the heart (QTcF) and the effectiveness of afatinib (BIBW 2992) in treating certain cancers. Cancers studied will include glioblastoma and cancers which have spread to the brain (metastases).

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients aged at least 18 years old.
2. Histologically or cytologically confirmed diagnosis of a solid malignant tumour, known to express EGFR/HER2 that is either refractory to standard therapies, or for which no standard treatment is available (including patients with brain metastases).
3. At least one tumor lesion that can accurately be measured by computed tomography (CT) or magnetic resonance imaging (MRI) in at least one dimension with longest diameter to be recorded as greater than or equal to 20 mm using conventional techniques or greater than or equal to 10 mm with spiral CT scan.
4. Life expectancy of at least 3 months.
5. Written informed consent that is consistent with ICH-GCP guidelines.
6. Eastern Cooperative Oncology Group (ECOG) performance score 0,1 or 2.
7. Patients must have recovered from any previous surgery.
8. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) for the duration of trial participation. Female patients with reproductive potential must have a negative serum pregnancy test within 7 days of trial enrolment. Breast feeding mothers will be excluded since these agents may be toxic to infants.

For patients with Glioma and brain metastases the following additional inclusion criteria should apply:

1. Histologically-confirmed WHO Grade IV malignant glioma at first episode of recurrence after prior combined chemo-radiotherapy. Patients with prior low-grade glioma are eligible if histological assessment demonstrates transformation to WHO Grade IV malignant glioma.
2. Bi-dimensionally measurable disease with a minimum measurement of 1 cm (10 mm) in one diameter on Gd MRI performed within 14 days prior to first treatment (Day 1).

Exclusion criteria:

Major exclusion criteria; 9. Radiotherapy within the past 2 weeks prior to treatment with the trial drug. 10. Chemo-, hormone- (other than megestrol acetate or steroids required for maintenance non-cancer therapy) or immunotherapy within the past 4 weeks before first drug administration.

11. Patients not completely recovered from any therapy-related toxicities from previous chemo-, hormone-, immuno-, or radiotherapies to CTC < Grade 1. Prior chemotherapy is allowed if completed at least 4 weeks prior to first trial treatment (6 weeks for mitomycin C or nitrosoureas) and the patient has recovered from the acute toxicities of that therapy.

12. Prior treatment with EGFR targeting therapies or treatment with EGFR- or HER2 inhibiting drugs within the past four weeks before start of therapy or concomitantly with this trial.

15. History of clinically significant or uncontrolled cardiac disease, including congestive heart failure, angina, myocardial infarction, arrhythmia, including New York Heart Association (NYHA) functional classification of 3.

16. Cardiac left ventricular function with resting ejection fraction < 50% measured by multigated blood pool imaging of the heart (MUGA scan) or Echocardiogram.

17. QTcF- interval > 470 ms at screening. 18. PR-interval > 230 ms at screening. 19. QRS-interval >120 ms at screening. 20. ST-segment and T/U-wave abnormalities at screening, as will be assessed by a cardiology specialist of a central lab.

21. Absolute neutrophil count (ANC) < 1,500/mm3. 22. Platelet count < 100,000 / mm3. 23. Bilirubin > 1.5 mg / dl (>26 micro mol / L, SI unit equivalent). Aspartate amino transferase (AST) or alanine amino transferase (ALT) > or equal to three times the upper limit of normal (if related to liver metastases > five times the upper limit of normal).

24. Serum creatinine > 1.5 times of the upper normal limit or calculated/measured creatinine clearance > or equal to 45 ml / min.

25. Patients with known Interstitial Lung Disease (ILD) For Patients with glioma and brain metastases additional exclusion criteria apply;

1. Patients with untreated or symptomatic brain metastases. Patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least four (4) weeks, no history of cerebral oedema or bleeding in the past four (4) weeks. Steroids will be allowed. Anti-epileptic therapy will be allowed if no changes are anticipated within the initial 14 days of treatment (QTC-evaluation).
2. Less than 4 weeks between radiotherapy and start of study treatment, unless new enhancing lesion outside of radiation field or radiologically progressive on two consecutive MRI scans at least four weeks apart or biopsy-proven recurrence.
3. Less than two weeks from surgical resection (one week from prior stereotactic biopsy) or major surgical procedure.
4. Less than two weeks after previous chemotherapy (6 weeks from nitrosureas).
5. Less than four weeks from prior treatment with bevacizumab.
6. Treatment with other investigational drugs; participation in another clinical study within the past 2 weeks before start of therapy or concomitantly with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- United Kingdom (4):
  - 1200.24.4403 Boehringer Ingelheim Investigational Site, Guildford
  - 1200.24.4402 Boehringer Ingelheim Investigational Site, London
  - 1200.24.4404 Boehringer Ingelheim Investigational Site, London
  - 1200.24.4401 Boehringer Ingelheim Investigational Site, Sutton

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Patients with tumours known to historically (over)express epidermal growth factor receptor (EGFR)/human epidermal growth factor receptor (HER) 2 with and without brain metastases, and patients with recurrent glioblastoma receiving an oral dose of Afatinib 50 mg once daily (qd)
Period: Overall Study
Arm/Group | All Patients
Started | 60 (Treated)
Completed | 0
Not Completed | 60
Not completed — Progressive disease | 41
Not completed — Other Adverse Event | 14
Not completed — Withdrawal by Subject | 2
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR)
Description: OR is defined as complete response and partial response (PR) and was assessed according to the Macdonald criteria for glioblastomas and brain metastases and according to Response Evaluation Criteria in Solid Tumours version 1.0 (RECIST) for solid tumours (excluding glioblastomas).
Time Frame: Tumour assessments were performed at screening, week 8, week 16, week 24, and every 8 weeks thereafter.
Population: Treated Set (TS). TS consisted of all patients who received at least one dose of trial medication.
Measure: Number; unit: Participants with OR
Arm/Group | All Patients
Number analyzed (Participants) | 60
Participants with OR | 1

2. Primary Outcome: Average Time-matched QT Corrected by the Fridericia Formula (QTcF) Change From Baseline to Day 14
Description: Average time-matched QT corrected by the Fridericia formula (QTcF) change from baseline to day 14 over 1 to 24 hours following administration of afatinib.
Time Frame: The day before the first drug dose (baseline) and the day 14. Electrocardiograms (ECG) were performed at time point 0 and 1 hour (h), 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 10 h, 24 h thereafter.
Population: All patients in TS who had at least 1 time-matched pair of QT measurements available from baseline and from Day 14 of treatment.
Measure: Mean (Standard Error); unit: ms
Arm/Group | All Patients
Number analyzed (Participants) | 49
ms | -0.3 (1.5)

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first treatment to the occurrence of tumour progression or death, whichever came first. It was assessed according to the Macdonald criteria for glioblastomas and brain metastases and according to RECIST for solid tumours (excluding glioblastomas) as well as by the investigators assessment. Median time results from unstratified Kaplan-Meier estimates.
Time Frame: Tumour assessments were performed at screening, week 8, week 16, week 24, and every 8 weeks thereafter.
Population: All patients from TS who progressed or died.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | All Patients
Number analyzed (Participants) | 53
weeks | 10.6 [7.4 to 15.0]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as time from start of treatment to death.
Time Frame: Tumour assessments were performed at screening, week 8, week 16, week 24, and every 8 weeks thereafter.
Population: TS.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | All Patients
Number analyzed (Participants) | 53
weeks | 39.6 [23.3 to NA]

5. Secondary Outcome: Disease Control
Description: Disease control was defined as CR, PR or stable disease (SD) and was assessed according to the Macdonald criteria for glioblastomas and brain metastases and according to RECIST for solid tumours (excluding glioblastomas).
Time Frame: Tumour assessments were performed at screening, week 8, week 16, week 24, and every 8 weeks thereafter.
Population: TS.
Measure: Number; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 60
Participants | 32

6. Secondary Outcome: Duration of Disease Control (DC)
Description: Duration of Disease control (DC). DC was defined as CR, PR or stable disease (SD) and was assessed according to the Macdonald criteria for glioblastomas and brain metastases and according to RECIST for solid tumours (excluding glioblastomas).
Time Frame: Tumour assessments were performed at screening, week 8, week 16, week 24, and every 8 weeks thereafter.
Population: TS.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | All Patients
Number analyzed (Participants) | 32
weeks | 15.3 [15.0 to 24.0]

7. Secondary Outcome: Patients With Notable Findings in QTcF on Day 14
Description: Notable findings are defined as a QTcF>500 ms or an increase in QTcF of >60ms.
Time Frame: Day 14
Population: All patients from TS with data for QTcF on day 14
Measure: Number; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 51
Participants | 1

8. Secondary Outcome: Patients With Clinically Relevant Findings in ECG on Day 14
Description: Patients with clinically relevant findings in Electrocardiogram data (ECG) on day 14.
Time Frame: Day 14
Population: All patients from TS with data for ECG on day 14
Measure: Number; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 51
Participants | 1

9. Secondary Outcome: Time-matched QTcF Changes From Baseline to Day 14 at Each Time-point
Description: Individual QTcF measurements at each time-point. Response was defined as the change from baseline. Analysis adjusted for baseline using a mixed model.
Time Frame: Baseline and day 14 (at 1, 2, 3, 4, 5, 6, 7, 10, 24 hours post-dose )
Population: All patients in TS who had at least 1 time-matched pair of QT measurements available from either Day1 or Day 14 of treatment.
Measure: Mean (Standard Error); unit: ms
Arm/Group | All Patients
Number analyzed (Participants) | 49
ms
  Time-point 1:00 h (N=48) | 1.6 (2.2)
  Time-point 2:00 h (N=48) | 1.2 (2.2)
  Time-point 3:00 h (N=49) | -2.1 (2.2)
  Time-point 4:00 h (N=49) | -2.5 (2.2)
  Time-point 5:00 h (N=49) | -2.3 (2.2)
  Time-point 6:00 h (N=49) | -0.4 (2.2)
  Time-point 7:00 h (N=48) | 0.2 (2.2)
  Time-point 10:00 h (N=49) | 0.2 (2.2)
  Time-point 24:00 h (N=48) | 0.6 (2.2)

10. Secondary Outcome: Average Time-matched QT Change From Baseline to Day 14
Description: Average time-matched QT change from baseline to day 14 over 1 to 24 hours following administration of afatinib.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ms
Arm/Group | All Patients
Number analyzed (Participants) | 49
ms | -0.4 (2.6)

11. Secondary Outcome: Patients With Notable Findings in QT on Day 14
Description: Number of Patients with notable findings in QT on day 14. Notable findings are defined as a QT>500 ms.
Time Frame: Day 14
Population: All patients from TS with data for QTcF on day 14
Measure: Number; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 51
Participants | 0

12. Secondary Outcome: Average Time-matched Heart Rate Change From Baseline to Day 14.
Description: Average time-matched heart rate change from baseline to day 14.
Time Frame: The day before the first drug dose (baseline) and the day 14.
Population: as for outcome 2
Measure: Mean (Standard Error); unit: bpm
Arm/Group | All Patients
Number analyzed (Participants) | 49
bpm | 0.1 (1.2)

13. Secondary Outcome: Highest CTC Grade for Adverse Events
Description: Highest Common Terminology Criteria (CTC) grade for adverse events
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Population: All patients from TS with adverse events
Measure: Number; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 60
Participants
  Grade 1 | 1
  Grade 2 | 19
  Grade 3 | 27
  Grade 4 | 4
  Grade 5 | 9

14. Secondary Outcome: Area Under Curve 0-24 Hours (AUC0-24) on Day 1
Description: AUC0-24 represents the area under the concentration curve of afatinib in plasma from 0 to 24 hours on Day 1.
Time Frame: 0.05 hours (h) before dosing and 1h, 2h, 3h, 4h, 5h, 6h,7h, 10h and 24h after dosing on Day 1
Population: TS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | All Patients
Number analyzed (Participants) | 56
ng*h/mL | 482 (55.6)

15. Secondary Outcome: Maximum Concentration (Cmax)
Description: Cmax represents the maximum measured concentration of afatinib in plasma on Day 1.
Time Frame: 0.05 hours (h) before dosing and 1h, 2h, 3h, 4h, 5h, 6h,7h, 10h and 24h after dosing on Day 1
Population: TS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | All Patients
Number analyzed (Participants) | 60
ng/mL | 44.7 (58.9)

16. Secondary Outcome: Time From Dosing to the Maximum Concentration (Tmax)
Description: tmax represents the time from dosing to the maximum concentration of afatinib in plasma on Day 1.
Time Frame: 0.05 hours (h) before dosing and 1h, 2h, 3h, 4h, 5h, 6h,7h, 10h and 24h after dosing on Day 1
Population: TS.
Measure: Median (Full Range); unit: hours
Arm/Group | All Patients
Number analyzed (Participants) | 60
hours | 3.06 [0.900 to 6.17]

17. Secondary Outcome: Area Under Curve of Afatinib Over a Uniform Dosing Interval Tau at Steady State (AUCtau,ss)
Description: AUCtau,ss represents the area under the concentration curve of afatinib in plasma over a uniform dosing interval tau (24h) at steady state (Day14).
Time Frame: 0.05 hours (h) before dosing and 1h, 2h, 3h, 4h, 5h, 6h,7h, 10h and 24h after dosing on Day 14
Population: TS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | All Patients
Number analyzed (Participants) | 44
ng*h/mL | 1250 (53.3)

18. Secondary Outcome: Maximum Concentration of Afatinib in Plasma at Steady State (Cmax,ss)
Description: Cmax,ss represents the maximum measured concentration of afatinib in plasma at steady state (Day 14).
Time Frame: 0.05 hours (h) before dosing and 1h, 2h, 3h, 4h, 5h, 6h,7h, 10h and 24h after dosing on Day 14
Population: TS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | All Patients
Number analyzed (Participants) | 44
ng/mL | 86.6 (55.2)

19. Secondary Outcome: Time From Dosing to the Maximum Concentration of Afatinib in Plasma at Steady State (Tmax,ss)
Description: tmax,ss represents the time from dosing to the maximum concentration of afatinib in plasma at steady state (Day 14).
Time Frame: 0.05 hours (h) before dosing and 1h, 2h, 3h, 4h, 5h, 6h,7h, 10h and 24h after dosing on Day 14
Population: Subset of TS, restricted to patients with adequate protocol compliance, i.e. patients without important protocol violations.
Measure: Median (Full Range); unit: hours
Arm/Group | All Patients
Number analyzed (Participants) | 44
hours | 3.07 [1.00 to 7.05]

20. Secondary Outcome: Accumulation Ratio of AUC Values (R_A,AUC)
Description: R_A,AUC represents the accumulation ratio of AUC values after multiple dose administration over a uniform dosing interval t between days 1 and 14
Time Frame: 0.05 hours (h) before dosing and 1h, 2h, 3h, 4h, 5h, 6h,7h, 10h and 24h after dosing on Day 1 and 14
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | All Patients
Number analyzed (Participants) | 42
ratio | 2.67 (53.4)

21. Secondary Outcome: Accumulation Ratio of AUC Values (R_A,Cmax)
Description: R_A,Cmax represents the accumulation ratio of Cmax values after multiple dose administration over a uniform dosing interval t between days 1 and 14
Time Frame: 0.05 hours (h) before dosing and 1h, 2h, 3h, 4h, 5h, 6h,7h, 10h and 24h after dosing on Day 1 and 14
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | All Patients
Number analyzed (Participants) | 44
ratio | 2.05 (58.5)

22. Secondary Outcome: Percentage Peak Trough Fluctuation (PTF)
Description: PTF represents the percentage peak trough fluctuation. PTF is defined as difference between maximum and minimum concentration at steady state divided by the average concentration multiplied with 100 to report as percentage.
Time Frame: 0.05 hours (h) before dosing and 1h, 2h, 3h, 4h, 5h, 6h,7h, 10h and 24h after dosing on Day 14
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of peak trough fluctuation
Arm/Group | All Patients
Number analyzed (Participants) | 44
percentage of peak trough fluctuation | 97.6 (37.8)

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 34/60
Other Adverse Events (participants affected / at risk) | 58/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=60)
Anaemia (Blood and lymphatic system disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Duodenal ulcer (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea/Vomiting (Gastrointestinal disorders) | 6
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 4
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Renal insufficency (Renal and urinary disorders) | 5
Urinary retention (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Rash/acne (Skin and subcutaneous tissue disorders) | 2
Ureteric obstruction (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=60)
Ocular effect (Eye disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 44
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 5
Nausea/Vomiting (Gastrointestinal disorders) | 28
Stomatitis (Gastrointestinal disorders) | 27
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 4
Pyrexia (General disorders) | 7
Lower respiratory tract infection (Infections and infestations) | 4
Nail effect (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 23
Dehydration (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Fatigue (Nervous system disorders) | 31
Headache (Nervous system disorders) | 4
Dysuria (Renal and urinary disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 8
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Rash/acne (Skin and subcutaneous tissue disorders) | 45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.